CLINICAL TRIAL: NCT00081458
Title: A Study of the Efficacy and Safety of Teduglutide in Subjects With Parenteral Nutrition-Dependent Short Bowel Syndrome
Brief Title: Safety and Efficacy Study of Teduglutide in Subjects With Short Bowel Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CL0600-004; 2004-000438-35 (EudraCT Number)
Record Dates: First submitted 2004-04-13; First posted 2004-04-14 (Estimated); Results first posted 2013-07-15 (Estimated); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Short Bowel Syndrome
Keywords: Short Bowel Syndrome; Parenteral Nutrition; SBS
MeSH Terms: conditions — Short Bowel Syndrome; Hyperphagia | interventions — teduglutide; ALX-0600

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- placebo (Placebo Comparator): Placebo injectable subcutaneously daily into the thigh or abdomen
  Interventions: Drug: Placebo
- 2 (Experimental): teduglutide 0.05 mg/kg/d
  Interventions: Drug: Teduglutide 0.05 mg/kg/d
- 3 (Experimental): teduglutide 0.1 mg/kg/d
  Interventions: Drug: Teduglutide 0.1 mg/kg/d

INTERVENTIONS:
Drug: Placebo — placebo injectable subcutaneously daily into thigh or abdomen
  Arms: placebo
Drug: Teduglutide 0.05 mg/kg/d — Teduglutide 0.05 mg/kg/d daily injectable subcutaneously into the thigh or abdomen
  Other Names: GATTEX
  Arms: 2
Drug: Teduglutide 0.1 mg/kg/d — Teduglutide 0.1 /g/kg/d daily injection subcutaneously into thigh or abdomen
  Other Names: GATTEX
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, tolerability, and pharmacokinetics (PK) of teduglutide compared with placebo in subjects with parenteral nutrition (PN)-dependent short bowel syndrome (SBS).

DETAILED DESCRIPTION:
Teduglutide is an analog of glucagon-like peptide 2 (GLP-2), a naturally occurring hormone that regulates the growth, proliferation, and maintenance of cells lining the gastrointestinal tract. Teduglutide has been shown in animal studies and previous human clinical trials to increase the size and number of these cells, thereby increasing the absorptive surface area of the intestines.

The multicenter, double-blind, international Phase III trial will randomly assign approximately 80 patients to receive daily subcutaneous injections of 0.05 milligrams or 0.10 milligrams of teduglutide per kilogram of body weight, or a placebo. Dosing will continue for a period of six months. The primary endpoint in the study is a reduction in the use of intravenous feeding, which is often required to sustain life in patients with SBS.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged 18 years of age or older at the time of signing the informed consent form (ICF)
* SBS as a result of major intestinal resection resulting in at least 12 months intravenous feeding
* Body weight must be less than 90 kg
* At baseline, subjects must require PN treatment to meet their caloric or electrolyte needs due to ongoing malabsorption at least 3 times weekly and to be on a stable PN regimen for 4 weeks before dosing
* Body mass index (BMI) 18 to 27 kg/m2
* Adequate hepatic and renal function

Exclusion Criteria:

* History of cancer or clinically significant lymphoproliferative disease with fewer than 5 years documented disease-free state
* History of alcohol or drug abuse (within previous year)
* Participation in a clinical study within 30 days prior to signing the ICF, or concurrent participation in any clinical study
* Clinically significant laboratory abnormalities at the time of randomization
* Previous use of teduglutide (ALX-0600)
* Prior use of native GLP-2 within 3 months of screening visit
* Hospital admission within 1 month prior to screening visit
* Pregnant or lactating women
* Any condition or circumstance, which in the investigator's opinion would put the subject at any undue risk, prevent completion of the study, or interfere with analysis of the study results.
* Presence of excluded disease: Radiation enteritis, Scleroderma, Celiac disease, Refractory/Tropical sprue, Pseudo-obstruction, Active inflammatory bowel disease (IBD), Pre-malignant/malignant change in colonoscopy biopsy or polypectomy, Surgery scheduled within the time frame of the study, Human immunodeficiency virus (HIV) positive test, Immunological disorders, Possible allergies to teduglutide or its constituents, Significant, active, uncontrolled, untreated systemic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2004-05-25 (Actual); Primary Completion 2007-07-06 (Actual); Study Completion 2007-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (32):
- United States (14):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Georgetown University, Washington D.C., District of Columbia
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern Center for Clinical Research, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Albany Medical Center, Albany, New York
  - Mount Sinai School of Medicine, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania - Penn Nursing, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
- l'Hôpital Erasme, Brussels, Belgium
- Canada (4):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
- Rigshospitalet, University of Copenhagen, Copenhagen, Denmark
- France (4):
  - Hôpital Claude-Huriez, Lille
  - Hôpital de la Croix-Rousse, Lyon
  - Hôpital Edouard Herriot, Lyon
  - Hôpital Beaujon, Paris
- Germany (3):
  - Charité University Hospital, Berlin
  - Charité-Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Frankfurt, Frankfurt
- Academic Medical Center, Amsterdam, Netherlands
- Poland (2):
  - Pracownia Żywienia Klinicznego, Olsztyn
  - Samodzielny Publiczny Szpital Kliniczny-Im.prof W.Orłowskiego CMKP, Warsaw
- United Kingdom (2):
  - Hope Hospital, Salford, Greater Manchester
  - St. Mark's Hospital, Harrow

REFERENCES:
- [Background] Dudrick SJ, Latifi R, Fosnocht DE. Management of the short-bowel syndrome. Surg Clin North Am. 1991 Jun;71(3):625-43. doi: 10.1016/s0039-6109(16)45438-1. PMID 1904648
- [Background] Rombeau JL, Rolandelli RH. Enteral and parenteral nutrition in patients with enteric fistulas and short bowel syndrome. Surg Clin North Am. 1987 Jun;67(3):551-71. doi: 10.1016/s0039-6109(16)44232-5. PMID 3109044
- [Background] Shanbhogue LK, Molenaar JC. Short bowel syndrome: metabolic and surgical management. Br J Surg. 1994 Apr;81(4):486-99. doi: 10.1002/bjs.1800810404. PMID 8205419
- [Background] Vanderhoof JA, Langnas AN. Short-bowel syndrome in children and adults. Gastroenterology. 1997 Nov;113(5):1767-78. doi: 10.1053/gast.1997.v113.pm9352883.
- [Result] Jeppesen PB, Gilroy R, Pertkiewicz M, Allard JP, Messing B, O'Keefe SJ. Randomised placebo-controlled trial of teduglutide in reducing parenteral nutrition and/or intravenous fluid requirements in patients with short bowel syndrome. Gut. 2011 Jul;60(7):902-14. doi: 10.1136/gut.2010.218271. Epub 2011 Feb 11. PMID 21317170
- [Derived] Fujioka K, Jeejeebhoy K, Pape UF, Li B, Youssef NN, Schneider SM. Patients With Short Bowel on Narcotics During 2 Randomized Trials Have Abdominal Complaints Independent of Teduglutide. JPEN J Parenter Enteral Nutr. 2017 Nov;41(8):1419-1422. doi: 10.1177/0148607116663481. Epub 2016 Aug 9. PMID 27507402

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject was screened 25May2004 and last subject evaluations were completed on 06Jul2007.
Pre-assignment Details: Patients underwent stabilization period for parenteral nutrition prior to randomization
Groups:
- Placebo: Placebo injected subcutaneously daily
- Teduglutide 0.05 mg/kg/d: teduglutide 0.05 mg/kg/d injected subcutaneously
- Teduglutide 0.1 mg/kg/d: teduglutide 0.1 mg/kg/d injected subcutaneously
Period: Overall Study
Arm/Group | Placebo | Teduglutide 0.05 mg/kg/d | Teduglutide 0.1 mg/kg/d
Started | 16 | 35 | 33
Received Treatment | 16 | 35 | 32 (1 subject was randomized but did not receive the study drug)
Completed | 15 | 27 | 29
Not Completed | 1 | 8 | 4
Not completed — Adverse Event | 1 | 5 | 2
Not completed — Withdrawal by Subject | 0 | 3 | 1
Not completed — Randomized but not dosed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: 84 subjects were initially randomized; however, one subject never received study therapy. As a result, the total participant who started flow period is 83.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Teduglutide 0.05 mg/kg/d | Teduglutide 0.1 mg/kg/d | Total
Number analyzed (Participants) | 16 | 35 | 32 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (15.1) | 47.1 (14.2) | 50.3 (14.0) | 48.8 (14.2)
Age, Customized [Count of Participants; unit: Participants]
  < 35 years | 3 | 7 | 5 | 15
  35-44 years | 2 | 5 | 4 | 11
  45 - 54 years | 3 | 12 | 10 | 25
  > 55 years | 8 | 11 | 13 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 18 | 19 | 46
  Male | 7 | 17 | 13 | 37
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 1 | 1 | 0 | 2
  Canada | 1 | 2 | 5 | 8
  Denmark | 2 | 3 | 3 | 8
  France | 2 | 5 | 2 | 9
  Germany | 0 | 0 | 2 | 2
  Netherlands | 0 | 4 | 1 | 5
  Poland | 3 | 6 | 8 | 17
  United Kingdom | 0 | 3 | 1 | 4
  United States | 7 | 11 | 10 | 28

OUTCOME MEASURES:

1. Primary Outcome: A Graded Response Score in Parenteral Nutrition (PN) Reduction
Description: The intensity of the response relied on a reduction from Baseline in weekly parenteral nutrition (PN) volume (minimum reduction of 20% and a maximum of 100%). Duration of the response incorporated responses at Weeks(Wk) 16-20 and at Wk20-24. Zero (0 - lowest) assigned if <20% reduction at Wk20-24 and reduction at Wk16-20 of < 20%, 20-39%, or >=40%. One (1) assigned if reduction of 20-39% at Wk20-24 but < 20% at Wk16-20. Two(2) assigned if reductions of 40-99% at Wk20-24 AND <20% at Wk16-20 OR 20-39% at Wk20-24 AND 20-39% at Wk16-20. Three (3) assigned if reductions of 100% at Wk20-24 AND <20% at Wk16-20 OR 40-99% at Wk20-24 AND 20-39% at Wk16-20 OR 20-39% at Wk20-24 AND >=40% at Wk16-20. Four (4) assigned if reductions of 100% at Wk20-24 AND 20-39% at Wk16-20 OR 40-99% at Wk20-24 AND >=40% at Wk16-20.
Time Frame: 6 months
Population: Intent to Treat (ITT) analysis using a stepdown procedure that was stopped if the 0.10 mg/kg dose was not significantly better than placebo.
Measure: Number; unit: participants
Arm/Group | Placebo | Teduglutide 0.05 mg/kg/d | Teduglutide 0.1 mg/kg/d
Number analyzed (Participants) | 16 | 35 | 32
participants
  0 (No Response) | 15 | 19 | 24
  1 | 0 | 6 | 2
  2 | 1 | 6 | 4
  4 | 0 | 2 | 2
  5 (No longer need PN) | 0 | 2 | 0
Statistical Analysis 1: Comparison: Placebo vs Teduglutide 0.05 mg/kg/d vs Teduglutide 0.1 mg/kg/d; Test type: Superiority or Other; p = 0.007, ANCOVA

2. Secondary Outcome: Number of Subjects Achieving Binary Response at Week 20, Maintained at Week 24
Description: An efficacy responder was defined as achieving at least a 20% reduction from Baseline to Week 20 and maintained at Week 24 in weekly actual PN infusion volume.
Time Frame: 6 months of treatment
Measure: Number; unit: participants
Groups:
- Placebo: Placebo injected subcutaneously daily into the thigh or abdomen
Arm/Group | Placebo | Teduglutide 0.05 mg/kg/d | Teduglutide 0.1 mg/kg/d
Number analyzed (Participants) | 16 | 35 | 32
participants
  Responder | 1 [0 to 18.1] | 16 [29.2 to 62.2] | 8 [10.0 to 40.0]
  Non-Responder | 15 [0 to 0] | 19 [0 to 0] | 24 [0 to 0]
Statistical Analysis 1: Comparison: Placebo vs Teduglutide 0.05 mg/kg/d vs Teduglutide 0.1 mg/kg/d; An efficacy responder was defined as achieving at least a 20% reduction from Baseline to Week 20 and maintained at Week 24 in weekly actual PN infusion volume; Test type: Superiority or Other; p = 0.005, ANCOVA

ADVERSE EVENTS:
Time Frame: 6 months
Description: A total of 84 subjects were randomized in this study; however, one subject did not receive study drug. Thus, the safety population consists of 83 subjects.
Arm/Group | Placebo | Teduglutide 0.05 mg/kg/d | Teduglutide 0.1 mg/kg/d
Serious Adverse Events (participants affected / at risk) | 5/16 | 13/35 | 11/32
Other Adverse Events (participants affected / at risk) | 15/16 | 33/35 | 31/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=16) | Teduglutide 0.05 mg/kg/d (N=35) | Teduglutide 0.1 mg/kg/d (N=32)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colonic stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Short-bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Catheter related complication (General disorders) | 3 (3) | 0 (0) | 3 (3)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (2) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Gallbladder perforation (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Catheter bacteraemia (Infections and infestations) | 1 (1) | 1 (2) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Catheter sepsis (Infections and infestations) | 1 (3) | 3 (10) | 4 (5)
Catheter site infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Fungemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (4) | 0 (0)
Device failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Eye Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Intestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Medical device complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Drug level increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral discitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Coma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Catheterization venous (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=16) | Teduglutide 0.05 mg/kg/d (N=35) | Teduglutide 0.1 mg/kg/d (N=32)
abdominal distension (Gastrointestinal disorders) | 0 (0) | 6 (7) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 7 (12) | 9 (11)
diahrrea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (4)
Nausea (Gastrointestinal disorders) | 4 (4) | 5 (7) | 10 (13)
Asthenia (General disorders) | 0 (0) | 3 (3) | 2 (2)
Catheter related complications (General disorders) | 3 (3) | 1 (1) | 3 (4)
Fatigue (General disorders) | 2 (2) | 1 (1) | 5 (7)
Injection site bruising (General disorders) | 0 (0) | 1 (1) | 7 (8)
Injection site erythema (General disorders) | 0 (0) | 1 (1) | 6 (6)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 4 (5)
Pain (General disorders) | 1 (1) | 0 (0) | 4 (4)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (8) | 6 (7)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 4 (5) | 2 (4)
Pyrexia (General disorders) | 1 (1) | 3 (3) | 3 (6)
Catheter sepsis (Infections and infestations) | 2 (4) | 4 (12) | 4 (5)
Catheter site infection (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 3 (3) | 4 (4)
Nasopharyngitis (Infections and infestations) | 2 (2) | 6 (9) | 5 (7)
Urinary tract infection (Infections and infestations) | 3 (3) | 3 (7) | 5 (6)
Intestinal stoma complications (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (4) | 3 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 1 (1) | 9 (29) | 7 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less